CLINICAL TRIAL: NCT06128135
Title: Identify the Prosthesis Users' Necessities Concerning Their Devices.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Federal University of Espirito Santo (Other)
Responsible Party: Sponsor
Other Study IDs: 202310261600
Record Dates: First submitted 2023-10-27; First posted 2023-11-13 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Upper Limb Amputation at the Hand

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prosthesis Users: 30 participants, aged between 18 and 60, will be part of the study. The users must have at least 6 months of experience using upper limb prostheses. They will be asked a 15-question survey about their upper limb prostheses.
  Interventions: Other: Technology acceptance questionnaire for prostheses users.
- Therapists: 10 therapists that have experience working with prostheses. They will be asked a 9-question survey about upper limb prostheses that they usually handle.
  Interventions: Other: Technology acceptance questionnaire for therapists
- Relatives: 30 of the prosthesis users' relatives who live with the person and see the daily difficulties of using the device. They will be asked a 9-question survey about the device that their relatives costume to use.
  Interventions: Other: Technology acceptance questionnaire for relatives of prostheses users.

INTERVENTIONS:
Other: Technology acceptance questionnaire for prostheses users. — One questionnaire, which is for prosthesis users, where will be 15 questions to identify what kind of activities the person uses the prosthesis, how much is the use time and what is the main problem with the device.
  Groups: Prosthesis Users
Other: Technology acceptance questionnaire for relatives of prostheses users. — One questionnaire, where there will be between 8 questions to analyze which device characteristics, they think cause major discomfort during the use and could be improved.
  Groups: Relatives
Other: Technology acceptance questionnaire for therapists — One questionnaire, where there will be between 9 questions to analyze which device characteristics, they think cause major discomfort during the use and could be improved.
  Groups: Therapists

SUMMARY:
Despite many advances in prosthesis development, there are still some areas that need to be improved. One of them is the weight of the devices which could cause muscular fatigue in long-term use of the prosthesis and even abandonment. This study aims to identify the desired improvements in prosthetic devices from the perspective of the users, therapists, and relatives. That would be done through two kinds of questionnaires about technology acceptance.

DETAILED DESCRIPTION:
The World Health Organization (WHO) estimates that around 1.3 billion people experience significant disability. One of the actual challenges is facilitating and breaking the barriers of persons with disabilities. Assistance technology supports inclusion and participation, principally for people with disabilities.

In Brazil, the DATASUS estimated that around 57802 amputations (one kind of disability) were performed in 2022. Prostheses are assistive devices that aim to mitigate the psychological impact of missing a member and help in activities of daily life (ADL). One kind of prosthesis is electrically powered, which uses electrical components to actuate the device and is commonly controlled by body signals such as surface electromyography (sEMG). Despite many advances in prosthesis development, some areas need to be improved such as weight, size, ergonomic design, etc. of the devices which could cause muscular fatigue in long-term use of the prosthesis and even abandonment.

This study aims to identify the aspects that cause major discomfort in upper limb prosthesis users. Also, recognize in which activities of daily life, the prosthesis is involved. That information will be used to improve the design of an upper limb prosthesis.

For the execution, two kinds of questionnaires about technology acceptance will be used. In the first questionnaire, which is for prosthesis users, there will be 15 questions to identify in what kind of activities the person uses the prosthesis, how much is the use time and what is the main problem with the device. In the second questionnaire, which is for the therapist and relatives, there will be 9 questions to analyze which device characteristics cause major discomfort during the use and could be improved.

ELIGIBILITY:
Inclusion Criteria:

* Prosthesis users with at least 6 months of device use.
* Therapists with experience in working with amputees.
* Relatives of the prosthesis users.

Exclusion Criteria:

-

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Inhabitants of Brazil, from the state of Espírito Santo. The participants are associated with the Crefes rehabilitation center.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients that have an unconformity with the weight of the device and which functional characteristics they would improve their devices | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Reabilitação Física do Espírito Santo, Vila Velha, Espírito Santo, Brazil

DOCUMENTS (2):
  • Study Protocol (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/35/NCT06128135/Prot_000.pdf
  • Informed Consent Form (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT06128135/ICF_001.pdf